CLINICAL TRIAL: NCT05692700
Title: THE EFFECT OF INHALED LAVENDER AND BERGAMOT OIL ON ANXIETY AND SLEEP QUALITY OF SURGICAL INTENSIVE CARE PATIENTS
Brief Title: The Effect of Inhaled Lavender and Bergamot Oil on Anxiety and Sleep Quality in Intensive Care Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, ÇAĞLA TOPRAK, specialist nurse, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: E-95961207-604.01.01-1535
Record Dates: First submitted 2022-12-16; First posted 2023-01-20 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2022-12

CONDITIONS: Patient Undergoing Surgery
Keywords: Intensive care unit,; sleep quality,; anxiety; aromatherapy,; lavender oil,; bergamot oil
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Anxiety Disorders | interventions — Aromatherapy

STUDY DESIGN:
Intervention Model Description: - Having pain, having smell problems, having systolic blood pressure below 100 mm Hg, having lung cancer, asthma and chronic obstructive pulmonary disease, allergic to known plants, flowers and related essential oils, using any medication for anxiety and sleep problems Lavender and bergamot oil were not administered to the patients by inhalation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Aromatherapy lavender group (Experimental): Stage 1: Patient information form, follow-up form, State Continuity Anxiety Scale, Richard-Campbell Sleep Scale were filled.Stage 2: On the second day of the surgery, at 20:00 in the evening, they were asked to inhale 2-3 drops of lavender essential oil, which was dripped onto the pillow pouches, at 21:00, and these bags were placed 10 cm away from the patient after 20 minutes. These bags were taken from the bedside of the patient at 08:00 in the morning.. Stage 3: Before the evening application, the patient follow-up form, State-Continuity Anxiety Scale, Richard Campbell Sleep Scale were filled and they were asked to inhale 2-3 drops of lavender essential oil, which was dropped on the pillow bags prepared at 20:00, and inhaled at 21:00. Afterwards, these sacs were placed 10 cm away from the patient. These sacs were taken from the bedside of the patient at 08:00 in the morning and the patient follow-up Form, State-Trait Anxiety Scale, Richards-Campbell Sleep Scale were filled
  Interventions: Other: aromatherapy
- Aromatherapy bergamot group (Experimental): Stage1:Patient information form, follow-up form, State Continuity Anxiety Scale, Richard Campbell Sleep Scale were filled. Stage 2:On the second day of the surgery, at 20:00 in the evening, they were asked to inhale 2-3 drops of bergamot essential oil, which was dripped onto the pillow pouches,at 21:00, and these bags were placed 10 cm away from the patient after 20 minutes. These bags were taken from the bedside of the patient at 08:00 in the morning.Stage 3:Before the evening application, the patient follow-up form, State-Continuity Anxiety Scale, Richard Campbell Sleep Scale were filled and they were asked to inhale 2-3 drops of bergamot essential oil, which was dropped on the pillow bags prepared at 20:00, and inhaled at 21:00. Afterwards, these sacs were placed 10 cm away from the patient.These sacs were taken from the bedside of the patient at 08:00 in the morning and the patient follow-up Form, State-Trait Anxiety Scale, Richards-Campbell Sleep Scale were filled.
  Interventions: Other: aromatherapy
- Plasebo group (Placebo Comparator): Stage 1:Patient identification form, follow-up form, State Continuity Anxiety Scale, Richard Campbell Sleep Scale were filled in.Stage2: 2-3 drops of distilled water dripped onto the prepared pillow bags at 21:00 on the second and third days of the surgery by inhalation. They were asked to breathe and after 20 minutes, these sacs were taken and placed 10 cm away from the patient.Stage 3:These sacs were taken from the bedside of the patient at 08:00 in the morning and the patient follow-up form, State-Trait Anxiety Scale, Richards Campbell Sleep Scale were filled again.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: aromatherapy — essential oil application by inhalation
  Arms: Aromatherapy bergamot group; Aromatherapy lavender group
Other: Placebo — Placebo essential oil
  Arms: Plasebo group

SUMMARY:
This study was carried out as a randomized controlled experimental study to determine the effect of inhaled lavender and bergamot oil on anxiety and sleep quality in patients hospitalized in the intensive care unit who had undergone surgical intervention.

The universe of the research; Patients who were hospitalized in an Intensive Care Unit in Istanbul between May 2021 and October 2021, and the sample consisted of patients who met the criteria for inclusion in the study. Fifty-four patients who agreed to participate in the study and met the inclusion criteria were included. Lavender oil or bergamot oil or distilled water was administered to the patients 2 evenings by inhalation.

DETAILED DESCRIPTION:
The universe of the research; Patients who were hospitalized in the Intensive Care Unit of a university hospital in Istanbul between May 2021 and October 2021, and the sample consisted of patients who met the inclusion criteria of the study. Data collection started after obtaining the ethics committee permission, institutional permission, and research permission from the Ministry of Health GETAT Clinical Research Department. A simple computer-assisted randomization method was used to distribute the groups homogeneously. Fifty-four patients who were hospitalized in the reanimation intensive care unit and accepted to participate in the study and met the inclusion criteria were included. The patients were randomly assigned to 3 groups of 18 people, each with distilled water, lavender oil, and bergamot oil. "Patient Information Form", "Patient Follow-up Form", "State-Trait Anxiety Inventory" and "Richard-Campbell Sleep Scale (RCUS)" were used to collect data.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old and under 70 years old.
* Staying in the intensive care unit for at least 3 nights after surgery.
* Ability to communicate ("Richmond Agitation Sedation Scale" +1, 0, -1 points).
* Glasgow coma scale score of 9 or higher.

Exclusion Criteria:

* Having pain.
* Having any problems with smelling.
* The need for mechanical ventilation.
* Systolic blood pressure below 100 mm Hg.
* Having lung cancer, asthma and chronic obstructive pulmonary disease.
* Having allergies to known plants, flowers and related essential oils.
* Using any medication for anxiety and sleep problems.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2021-05-02 (Actual); Primary Completion 2021-10-20 (Actual); Study Completion 2021-11-03 (Actual)

PRIMARY OUTCOMES:
Insomnia in intensive care patients who have undergone surgery assessed by Richards-Campbell Sleep Scale | 1 year
  Richards-Campbell Sleep Scale In 1987, Richards K developed the Richard-Campbell Sleep Scale. It is used to evaluate sleep quality in patients and patients in the intensive care unit. The Richards-Campbell Sleep Scale evaluates sleep depth, time to fall asleep and number of awakenings, as well as sleep efficiency and quality with 6 questions. The sixth question was adapted to assess perceived night noise. The first 5 questions are taken into the calculation of the score, the score of the 6th question is not added. It is scored on a visual analog scale ranging from 0 mm to 100 mm, and low scores (0-25 points) represent poor sleep and higher scores (76-100 points) represent good sleep. The mean score of the five items is known as the total score and represents the overall perception of sleep.
Insomnia in intensive care patients who have undergone surgery assessed by State-Trait Anxiety Scale | 1 year
  State-Trait Anxiety Scale It is a scale used to evaluate the status, continuity and anxiety of patients. It is widely used in hospitals and clinics. The scale is in the form of two separate scales and consists of a total of forty items.
  The total score calculated from the two scales varies between 80 and 20. The higher the total anxiety score, the higher the anxiety level, and the lower the anxiety level, the lower the anxiety level.

CONTACTS AND LOCATIONS:
Locations (1):
- Çağla, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Cho MY, Min ES, Hur MH, Lee MS. Effects of aromatherapy on the anxiety, vital signs, and sleep quality of percutaneous coronary intervention patients in intensive care units. Evid Based Complement Alternat Med. 2013;2013:381381. doi: 10.1155/2013/381381. Epub 2013 Feb 17. PMID 23476690
- [Background] Muz G, Tasci S. Effect of aromatherapy via inhalation on the sleep quality and fatigue level in people undergoing hemodialysis. Appl Nurs Res. 2017 Oct;37:28-35. doi: 10.1016/j.apnr.2017.07.004. Epub 2017 Aug 1. PMID 28985917
- [Result] Chen ML, Chen YE, Lee HF. The Effect of Bergamot Essential Oil Aromatherapy on Improving Depressive Mood and Sleep Quality in Postpartum Women: A Randomized Controlled Trial. J Nurs Res. 2022 Apr 1;30(2):e201. doi: 10.1097/jnr.0000000000000459. PMID 34690334